CLINICAL TRIAL: NCT05088616
Title: Community Partnered Medical Nutrition Intervention for Native Americans Living with Diabetes
Brief Title: Native American Diabetes Project
Acronym: NADP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped primarily due to challenges recruiting and retaining participants. The investigators repeatedly tried to address this issue but still faced major challenges. Follow-up research was done to explore this challenge further.
Sponsor: University of Southern California (Other)
Collaborators: Project Angel Food (Unknown); United American Indian Involvement, Inc. (Unknown)
Responsible Party: Principal Investigator, Claradina Soto, Assistant Professor, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UP-20-01441
Record Dates: First submitted 2021-10-08; First posted 2021-10-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Diabetes; Diabete Type 2; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Type 1; Diabetes Mellitus
Keywords: American Indian; Alaska Native; Native American; Education; Wellness program; Meals; Nutrition; Classes; Tribal; Indigenous; Native; Social interaction; Diabetes; Blood sugar; Buddy; Urban Indian; Urban; online classes; virtual classes; Los Angeles; AIAN; Los Angeles County; A1c; blood; clinic; diabetes education; public health; social; social isolation; isolation; behavior; behavioral; culture; cultural connectedness; connection; well-being; population; population health; adults; urban population; race; chronic disease; food; healthy food; patient education; North America; California; Southern California; Pacific States; United States; ethnic and racial minorities; Indians, North American; Indigenous peoples; endocrine system diseases; diabetes mellitus; sugar; diet; meal delivery; early termination of clinical trials; surveys; Zoom; labs; blood test
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Social Isolation; Behavior; Chronic Disease; Endocrine System Diseases

STUDY DESIGN:
Intervention Model Description: All participants receive the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Virtual Diabetes Wellness Classes and Medically Tailored Meals (Experimental): All participants will receive the same intervention: four weeks of virtual diabetes wellness classes and 12 weeks of medically tailored meals. Additionally, participants will be paired with one to two "buddies" to provide support to each other.
  Interventions: Behavioral: Virtual Diabetes Wellness Classes and Medically Tailored Meals

INTERVENTIONS:
Behavioral: Virtual Diabetes Wellness Classes and Medically Tailored Meals — Four weeks of virtual diabetes wellness classes and 12 weeks of medically tailored meals.

SUMMARY:
This research study is for American Indian and Alaska Native (AIAN) people with diabetes in Los Angeles County, California. Participants (people who join the study) are signed up for a program that includes healthy meals, online diabetes classes, and social support.

This study aims to answer the following question:

Can this program (the meals, classes, and social support) have health and well-being benefits for participants, like lower blood sugar levels and less social isolation?

Participants are asked to fill out surveys and go to three clinic visits. Participants do not have to pay for the clinic visits or any other parts of the study.

DETAILED DESCRIPTION:
Diabetes in the American Indian and Alaska Native (AIAN) population is a public health crisis. AIAN have the highest diabetes prevalence rates when compared to other racial and ethnic populations in the United States. According to the Centers for Disease Control and Prevention, 14.7% of AIAN adults compared to 7.5% of non-Hispanic Whites have been diagnosed with diabetes. In California (CA), those who self-identify as having CA Tribal heritage are twice as likely than individuals from tribes outside of CA to be diagnosed with diabetes (31% versus 16%). Significant disparities also exist in diabetes-related outcomes. Compared to the general population, AIANs are 2.3 times more likely to die from diabetes, and the incidence of diabetes-related kidney failure among AIANs is 2.0 times higher. Cardiovascular disease among AIANs with diabetes may be 3-8 times higher than those AIAN without diabetes.

The diabetes crisis among AIAN is best addressed using a holistic approach. Aside from addressing the impact of diabetes on several physical health outcomes, best practices also include addressing the impact of trauma and mental and emotional health, providing robust patient education, and addressing structural barriers such as food insecurity, lack of access to healthy food, living in poverty, limited social support, and lack of access to health care, especially that which is culturally responsive.

Given the disproportionate rates of diabetes and diabetes-related outcomes among AIANs, this is the perfect opportunity to provide a culturally tailored health promotion intervention among the largest urban AIAN population in the U.S.; approximately 171,163 AIANs reside in Los Angeles County.

The goal of this pilot study was originally to reach up to 312 Native Americans with diabetes (later reduced, aiming for 150) to participate in an intervention to lower blood sugar and feelings of social isolation. The intervention will include 12 weeks of diabetes-friendly, medically tailored meals, and four weeks of virtual diabetes wellness classes. Each participant will be part of a 180-day cohort, during which participants will complete surveys and attend three clinic visits.

ELIGIBILITY:
Inclusion Criteria:

1. Reside in Los Angeles County,
2. 18 years and older,
3. Diabetic
4. Identify as American Indian or Alaska Native,
5. Have freezer space for 14 meals (about the size of two shoe boxes),
6. Ability to attend virtual classes via Zoom,
7. Ability to complete electronic surveys distributed by email,
8. Ability to commit to attending at least five of the six initial classes and meetings,
9. Ability to commit to making personal arrangements to attend three study clinic visits during weekday, daytime hours, and
10. Ability to consent to study activities, attend classes, and complete surveys all in English.

Exclusion Criteria:

1. Pregnancy,
2. Food allergies,
3. Serious non-allergic reactions to foods, and
4. Unable or unwilling to eat study meals (considering the limited accommodations available).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Change in A1c (from baseline to 90 days and 180 days) | Baseline, 90 days, and 180 days

SECONDARY OUTCOMES:
Change in blood pressure (from baseline to 90 days and 180 days) | Baseline, 90 days, and 180 days
Change in BMI (using weight and height) (from baseline to 90 days and 180 days) | Baseline, 90 days, and 180 days
Change in social isolation (using loneliness measure survey questions) (from baseline to 90 days and 180 days) | Baseline, 90 days, and 180 days
Change in level of diabetes distress (using diabetes distress scale survey responses) (from baseline to 90 days and 180 days) | Baseline, 90 days, and 180 days
Change in identity and level of cultural connectedness (using part of Multigroup Ethnic Identity Measure survey questions) (from baseline to 90 days and 180 days) | Baseline, 90 days, and 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Claradina Soto, PhD, MPH, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
While we understand the value of data sharing, research with Native American communities is particularly sensitive due to data sovereignty and past abuses, including the use of Native people's data for purposes the people didn't know about or agree to, sometimes causing harm to the community. Our informed consent states that even deidentified participant data will not be used or distributed for further studies. We made this choice out of respect for the data considerations here and also to ensure potential participants feel as comfortable as possible when participating, as recruitment can already be challenging.

REFERENCES:
- [Background] Centers for Disease Control and Prevention. (2020). National diabetes statistics report. https://www.cdc.gov/diabetes/data/statistics-report/index.html
- [Background] Garcia AN, Castro MC, Sanchez JP. Social and Structural Determinants of Urban American Indian and Alaska Native Health: A Case Study in Los Angeles. MedEdPORTAL. 2019 May 15;15:10825. doi: 10.15766/mep_2374-8265.10825. PMID 31161137
- [Background] Office of Disease Prevention and Health Promotion, n.d. Diabetes. Healthy people 2020. U.S. Department of Health and Human Services. https://www.healthypeople.gov/2020/data-search/Search-the-Data?topic-area=3514
- [Background] UCLA Center for Health Policy Research. (2017). American Indian and Alaska Native diabetes: critical information for researchers and policy-makers [Fact sheet]. https://healthpolicy.ucla.edu/publications/Documents/PDF/AIANDiabetesmay2012.pdf